CLINICAL TRIAL: NCT03592342
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Clinical Study to Assess the Safety and Efficacy of Three Doses of Clobetasol Propionate When Administered Intra-orally Twice Daily in Patients With Oral Lichen Planus (OLP) Using Rivelin®-CLO Patches
Brief Title: Intra-oral Treatment of OLP With Rivelin®-CLO Patches
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dermtreat (Industry)
Collaborators: Proinnovera GmbH (Industry); X-act Cologne Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DT-001-R-004
Record Dates: First submitted 2018-06-19; First posted 2018-07-19 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Oral Lichen Planus
Keywords: Patch; Rivelin-Clo Patch; Oral Lichen Planus; Ulcerative; Erythematous; OLP; OLPClinROM; OLPSSM
MeSH Terms: conditions — Lichen Planus, Oral; Ulcer | interventions — Clobetasol

STUDY DESIGN:
Intervention Model Description: Randomization will be 1:1:1:1 to 1 of the 4 parallel arms (3 active and 1 placebo) and patients will be stratified according to number of patches needed (1-3 and 4-6).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All 4 interventions will be similar in appearance and be allocated by use of a blinded kit number (each kit contains drug for 1 week).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Rivelin® plain patches (Placebo Comparator): Dosing is two times per day (morning and evening) with Rivelin® plain patches (placebo).
  Interventions: Drug: Clobetasol Propionate
- Rivelin®-CLO patch 1µg (Experimental): Dosing is two times per day (morning and evening) with Rivelin®-CLO patch 1µg Clobetasol propionate per patch.
  Interventions: Drug: Clobetasol Propionate
- Rivelin®-CLO patch 5µg (Experimental): Dosing is two times per day (morning and evening) with Rivelin®-CLO patch 5µg Clobetasol propionate per patch.
  Interventions: Drug: Clobetasol Propionate
- Rivelin®-CLO patch 20µg (Experimental): Dosing is two times per day (morning and evening) with Rivelin®-CLO patch 20µg Clobetasol propionate per patch.
  Interventions: Drug: Clobetasol Propionate

INTERVENTIONS:
Drug: Clobetasol Propionate — Rivelin® patch is a two-layer patch comprised of a muco-adhesive, drug-delivery layer and a protective layer.

SUMMARY:
Participants with symptomatic Oral Lichen Planus lesions will be treated with Rivelin® patches containing either 0, 1, 5, or 20 μg clobetasol per patch. Each participant will apply up to 6 patches twice daily for 4 weeks.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled, parallel group clinical study with 3 active dose arms (Rivelin®-CLO patches) and one placebo arm (Rivelin® plain patch). Up to 6 Rivelin® patches will be applied to symptomatic ulcerative and symptomatic erythematous OLP lesions.

After screening (visit 1, day -14 to day -7), patients who have signed the informed consent form and who are fulfilling the inclusion criteria and none of the exclusion criteria will be randomized at baseline (visit 2, day 1) to one of the four treatment arms in a double-blinded fashion.

* Arm A: Rivelin® plain patch (Placebo)
* Arm B: Rivelin®-CLO 1 μg/patch
* Arm C: Rivelin®-CLO 5 μg/patch
* Arm D: Rivelin®-CLO 20 μg/patch Randomization will be 1:1:1:1 and patients will be stratified according to number of patches needed (1-3 and 4-6).

The screening phase ranges between 7 and 14 days, i.e. that the screening visit (visit 1) needs to be performed 7 days prior to baseline at latest. For visits 3 (day 8), 4 (day 15), 5 (day 22), and 6 (day 29) a visit window of +/- 2 days will be allowed. Visit 7 will be defined as visit 6 + 14 days, with a visit window of +/- 3 days.

Randomized patients will enter a 28-days (4-weeks) treatment period. Dosing is two times per day (morning and evening) with patches applied directly on OLP lesions as instructed by a clinician or delegated site staff. Patients will record symptoms and adhesion time in daily diaries by using an electronic diary (eDiary).

During the treatment period, the treating physician or dentist will perform an assessment of the disease status on a weekly basis. A final examination of disease status will be performed at the follow-up visit (visit 7), 14 days after the end of treatment.

Other treatments of symptomatic OLP lesions during the study are prohibited. Only rescue analgesics determined by the investigator at study entry on a patient specific basis are allowed to be taken, in case that OLP associated symptoms like pain cannot be managed by the sole use of the patches. All doses of rescue analgesics will be recorded by the patient in the eDiary.

If the patients' condition is worsening (at the discretion of the investigator) and if associated symptoms cannot longer be managed acceptably by the additional use of rescue analgesics, i.e. if there is the need to start any other OLP treatment, IMP treatment for that patient should be discontinued prematurely and patient should be withdrawn from the study.

At visit 3 (day 8), a blood sample will be drawn to measure the blood plasma concentration of clobetasol and to determine the morning serum cortisol level (between 7 and 9 AM).

All patients will have a follow-up visit that will be performed 2 weeks after the EoT/ET visit (visit 6).

Safety data (by means of AE documentation including fungal infections and SAE reporting) will be closely monitored by an independent Data and Safety Monitoring Board (DSMB). DSMB will advise the Sponsor of any potential risk for the safeguard of patients.

ELIGIBILITY:
Inclusion Criteria:

* OLP patients with at least one visible and measurable symptomatic ulcerative OLP lesion, assessable via OLP Clinician Reported Outcome Measure (OLPClinROM).
* Diagnosis of LP histologically confirmed by result of either an existing clinically relevant biopsi or a new clinically representative biopsy at first screening visit (i.e. a biopsy report either indicative of OLP, LP or indicative of lichenoid inflammation will be sufficient).
* Patients aged ≥ 18 years.
* Patients practicing daily oral hygiene (by tooth brushing and/or mouth rinse) and willing to maintain at least their routine oral hygiene procedure during study participation.
* Willingness to keep already used permitted concomitant medication, food supplements (e.g. probiotics) or herbals, which might have in the discretion of the investigator a potential influence on OLP, on a stable basis during the study.

Exclusion Criteria:

* Patients requiring more than 6 patches (corresponding to an area of approximately 3 cm2 per patch) to cover symptomatic ulcerative and erythematous OLP lesions at baseline visit.
* Ongoing active visible fungal, bacterial or viral infection of oral mucosa, including ongoing treatment of those at baseline.
* Patient with any un-healed oral surgery (including recent diagnostic biopsies, if applicable) or oral laser therapeutic wound(s) at baseline visit.
* Any of the following systemic treatments prior to baseline visit and throughout the study:

  * Protease inhibitors used for the treatment of HIV (e.g. atazanavir, idinavir, nelfinavir, etc.): 1 week
  * Corticosteroids (i.v., intra articular, intra-lesional): 4 weeks
  * Antimycotics: 4 weeks The following systemic treatments are allowed, if on stable dose for a defined period of time to baseline and throughout the study.
  * Antibiotics: 4 weeks
  * Corticosteroids (oral, rectal, inhalative) washout/stable with maxinum dose of 10 mg daily prednisolone or equivalent for 4 weeks.
  * Retinoids: 12 weeks
  * Immunosuppressive drugs (e.g. azathioprine, cyclosporine, mycophenolate mofetil, or biologics): 12 weeks
* Any of the following topical treatments used in the oral cavity prior to baseline visit:

  * Corticosteroids: 2 weeks
  * Antibiotics: 2 weeks
  * Cyclosporine: 2 weeks
  * Tacrolimus, pimecrolimus: 2 weeks
  * Antimycotics: 2 weeks
  * Retinoids: 4 weeks
* Phototherapy in oral cavity prior to baseline visit: UVB, PUVA.
* Current participation in another clinical study and/or having received treatment with any non-marketed / investigational medicinal product (drug substance or medical device) within 4 weeks prior to screening.
* Known or suspected intolerance/hypersensitivity/resistance to clobetasol propionate or any component of the investigational medicinal product.
* Any history of squamous cell carcinoma (even if resected), as well as history of other non-squamous cell carcinoma (e.g. sarcoma, salivary gland tumors) that have been managed with radiation or chemotherapy.
* History of cancer (except resected cutaneous basal cell carcinoma and except in situ cervical cancer) unless it can be documented that the patient has been in a disease-free state for at least 5 years, or at least 2 years in a disease-free state for low-grade cancers. In case of clinical suspicion of malignancy in the oral cavity, a patient can only be included after an excluding biopsy.
* Professional dental cleaning within 2 weeks prior to baseline and unwillingness to refrain from professional dental cleaning during study conduct.
* Close affiliation with the investigator (e.g. a close relative) or persons working at the study sites or patient who is an employee of the Sponsor's company.
* Pregnant, confirmed by a positive pregnancy test, or nursing (lactating) women, or women of childbearing potential (WOCP) planning to become pregnant or WOCP not using or willing to continue to use a defined highly effective method of contraception throughout the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-06-28 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Change in ulcer area | 4 weeks
  The change will be calculated from baseline to end of trial

SECONDARY OUTCOMES:
Change in lesion area | 4 weeks
  The change will be calculated from baseline to end of trial
Change in 5-point erythema score | 4 weeks
  The change will be calculated from baseline to end of trial using a 5-point erythema score (assessed as no redness (0) or very severe redness (4))
Change in Clinical global impression score | 4 weeks
  The change will be calculated from baseline to end of trial using the Clinical Global Impression Score assessed on a 5-point rating scale ranging between no disease (0) and very severe disease (4)
Change in OLPSSM total score (item #1 to #7) | 4 weeks
  The change will be calculated from baseline to end of trial. The OLPSSM (OLP Symptom Severity Measure) is a recently developed questionnaire, which serves for the patient to assess his/her specific OLP symptoms. This questionnaire consists of overall 12 items, to be assessed at different time points. Most items should be completed on a daily basis (in the evening). These items will be assessed as part of the patient's eDiary
Change in individual diary symptom scores (item #1 to #7 of the OLPSSM) | 4 weeks
  The change will be calculated from baseline to end of trial. The OLPSSM (OLP Symptom Severity Measure) is a recently developed questionnaire, which serves for the patient to assess his/her specific OLP symptoms. This questionnaire consists of overall 12 items, to be assessed at different time points. Most items should be completed on a daily basis (in the evening). These items will be assessed as part of the patient's eDiary.
Change in worst symptoms at anatomical sites | 4 weeks
  The change will be calculated from baseline to end of trial
The proportion of positive outcomes (score 0 or 1) on each of the 11 questions in the Patch Sensation Questionnaire | 2 weeks
  The patient will assess the sensation of wearing the Rivelin® patches by answering 11 questions (the Patch sensation questionnaire) according to 5-point rating scales (ranging between 0 [most positive response] and 4 [most negative response]).The Patch Sensation Questionnaire will be completed during the clinic visit at baseline (visit 2) after first patch application and at visit 4 (2 weeks).
The proportion of patients with successful (>=80% of days on treatment) patch applications | 4 weeks
  Defined as an adhesion time more than 30 minutes during the 4 weeks treatment
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | 4 weeks
  Frequency and intensity of adverse events (AEs) reported during the study

CONTACTS AND LOCATIONS:
Overall Officials: Lars Siim Madsen, PhD, Study Chair — Dermtreat; Michael Brennan, DDS, Principal Investigator — Carolinas Healthcare System, Dept. of Oral Medicine
Locations (27):
- United States (14):
  - QWay Research, Hialeah, Florida
  - Vitae Research Center, LLC, Miami, Florida
  - Valencia Medical & Research Center, Miami, Florida
  - The Dental College of Georgia, Augusta, Georgia
  - Tufts University, School of Dental Medicine, Boston, Massachusetts
  - Brigham and Women's Hospital, Division of Oral Medicine and Dentistry, Boston, Massachusetts
  - NYU College of Dentistry, Bluestone Center for Clinical Research, New York, New York
  - UNC Dermatology and Skin Cancer Center, Chapel Hill, North Carolina
  - Carolinas Center for Oral Health, Charlotte, North Carolina
  - University of Pennsylvania Health System, Dept. Oral amd Maxillofacial Surgery, Philadelphia, Pennsylvania
  - Texas A&M University (TAMU), College of Dentistry, Dallas, Texas
  - UT Southwestern Medical Center Department of Surgery, Dallas, Texas
  - ENT Associates of Texas, Frisco, Texas
  - The Oral and Facial Surgery Center, Clearfield, Utah
- Canada (2):
  - Kaye Edmonton Clinic, Edmonton, Alberta
  - Health Sciences North, North East Cancer Center, Greater Sudbury, Ontario
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - University of Copenhagen Department of Odontology, Copenhagen
- LMU München, Klinik und Poliklinik für Dermatologie und Allergologie, Munich, Germany
- Cork University Dental School and Hospital, Cork, Ireland
- United Kingdom (7):
  - School of Dental Sciences Newcastel Upon Tyne, Newcastle upon Tyne, Newcastel
  - Edinburgh Dental Institute, Edinburgh
  - University of Glasgow Dental School, Glasgow
  - Leeds Dental Institute, Leeds
  - King´s College London Dental Institute, Oral Clinical Research Unit, London
  - University College London and University College London Hospitals Trust, London
  - University of Sheffield, School of Clinical Dentistry, Sheffield

IPD SHARING:
Plan to Share IPD: Undecided